CLINICAL TRIAL: NCT01961232
Title: Examination of Trans-pulmonary Biomarkers in Pulmonary Hypertension: a Potential Step Towards Personalized Therapy
Brief Title: Trans-pulmonary Biomarkers in Pulmonary Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Ken Monahan, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: IRB090650
Record Dates: First submitted 2013-09-19; First posted 2013-10-11 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; biomarker; cardiac; circulation; heart disease; lung disease
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pulmonary Hypertension & WHO group I: Participants with Pulmonary Hypertension with a WHO classification group I and are scheduled to have a right heart catheterization.
- Pulmonary Hypertension & WHO group II: Participants with Pulmonary Hypertension with a WHO classification group II and are scheduled to have a right heart catheterization.
- Without Pulmonary Hypertension: Participants without Pulmonary Hypertension
- Connective Tissue Disease: Participants without PH, but with connective tissue disease

SUMMARY:
The investigators are testing whether the addition of Pulmonary Hypertension-related biomarkers, measured across the pulmonary circulation, to the standard hemodynamic evaluation for Pulmonary Hypertension will lead to more informed choices of Pulmonary Hypertension therapy and improved patient outcomes.

DETAILED DESCRIPTION:
Eligible participants with known or suspected Pulmonary Hypertension undergoing a clinically indicated right heart catheterization may be enrolled. Clinical data and blood samples will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Undergoing RHC for PH evaluation

Exclusion Criteria:

* Anemia defined as Hgb < 10 g/dL and HCT < 30
* Pregnancy at the time of RHC (as assessed by urine or serum pregnancy test on the day of the procedure)
* Left ventricular ejection fraction ≤ 40%
* Atrial fibrillation at the time of RHC (as defined by telemetry monitoring or EKG on the day of the procedure)
* IPF, CTEPH, COPD/OSA as the dominant etiology of PH
* Patient is currently taking PH medication or long-acting nitrates at the time of their RHC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary Vascular Clinic
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Differences in Pulmonary Hypertension biomarkers in patients evaluated for Pulmonary Hypertension | At baseline

SECONDARY OUTCOMES:
Vasodilator-induced changes in Pulmonary Vascular Resistance (PVR) | At baseline
Vasodilator-induced changes in Pulmonary Hypertension biomarkers | At baseline

OTHER OUTCOMES:
Differences between Pulmonary Hypertension-related biomarkers in pulmonary circulation and peripheral-venous circulation | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ken Monahan, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Monahan K, Scott TA, Su YR, Lenneman CG, Zhao DX, Robbins IM, Hemnes AR. Reproducibility of intracardiac and transpulmonary biomarkers in the evaluation of pulmonary hypertension. Pulm Circ. 2013 Apr;3(2):345-9. doi: 10.4103/2045-8932.114762. PMID 24015334